CLINICAL TRIAL: NCT00590655
Title: Effect of Maintenance Programme on the Long Term Weight Reduction in Severely Obese Patients. A Randomized Controlled Trial
Brief Title: Maintenance Programme After Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Finnish Medical Foundation (Network)
Responsible Party: Tuula Pekkarinen, Peijas Hospital, Department of Internal medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 231410; Finnish Medical Foundation
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Last update posted 2008-01-10 (Estimated); Status verified 2007-12

CONDITIONS: Weight Loss; Morbid Obesity
Keywords: maintenance therapy
MeSH Terms: conditions — Weight Loss; Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): Treatment B includes a four month weight loss programme (10 weeks on a VLED and 17 weeks behavior modification visits). Treatment lasts 17 weeks and after that there will be one and two year control visits including weighing and questionnaires for eating behavior and quality of life.
  Interventions: Behavioral: weight loss programme
- 1 (Experimental): Treatment includes a four month weight loss programme (10 weeks on a VLED and 17 weeks behavior modification visits). After that a maintenance programme starts with monthly sessions for one year. Weight loss, quality of life, and eating behavior will be assessed at the end of the maintenance program and one year later.
  Interventions: Behavioral: weight loss programme with maintenance programme

INTERVENTIONS:
Behavioral: weight loss programme with maintenance programme — After usual weight loss treatment, there will be a one-year maintenance programme with monthly visits.
  Arms: 1
Behavioral: weight loss programme
  Arms: 2

SUMMARY:
The aim of this study is to compare a weight reduction programme with and without a maintenance programme in patients with severe obesity.

ELIGIBILITY:
Inclusion Criteria:

* BMI 35 kg/m2 or more
* Age 18-65 years

Exclusion Criteria:

* Type 1 diabetes
* Major alcohol problem
* Acute psychic disease, eating behavior, pregnancy, severe disease (cancer, unstable coronary disease, severe liver or kidney disease), or the patient has been in this treatment within the past 5 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2002-08; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
weight result | 2 years after weight loss phase

SECONDARY OUTCOMES:
quality of life and eating behavior | 2 years after active weight loss

CONTACTS AND LOCATIONS:
Locations (1):
- Peijas Hospital, Vantaa, Finland

REFERENCES:
- [Derived] Pekkarinen T, Kaukua J, Mustajoki P. Long-term weight maintenance after a 17-week weight loss intervention with or without a one-year maintenance program: a randomized controlled trial. J Obes. 2015;2015:651460. doi: 10.1155/2015/651460. Epub 2015 Mar 30. PMID 25918644